CLINICAL TRIAL: NCT03448380
Title: FreeStyle Libre Flash Glucose Monitoring System Post Approval Study
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-PMS-17168-001
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SMBG and FreeStyle Libre: During the intervention phase, subjects will use FreeStyle Libre Flash Glucose Monitoring System for 6 months to managed their diabetes.
  Interventions: Device: FreeStyle Libre Flash Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitoring System — Subjects will utilize capillary SMBG for managing diabetes for 6 months (control phase) followed by diabetes management using FreeStyle Libre for 6 months (intervention phase).

SUMMARY:
This is a prospective, multi-center, non-randomized, single-arm, post-approval study of the FreeStyle Libre Flash Glucose Monitoring System intended to characterize the safety of the Libre Flash Glucose Monitoring System when used in people with diabetes.

DETAILED DESCRIPTION:
Up to 920 adult subjects, aged 18 years and older with type 1 or type 2 diabetes, who require daily blood glucose monitoring to manage their diabetes, will be enrolled to obtain at least 736 subjects who complete the final visit. Subjects will utilize capillary SMBG for managing diabetes for 6 months (control phase) followed by diabetes management using FreeStyle Libre for 6 months (intervention phase). Subjects will maintain a diary/log book of Adverse Events during each phase. Assessment of Adverse Events will occur via self reporting at each monthly visit and/or phone call.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject must have a diagnosis of type 1 or type 2 diabetes mellitus.
* Subject is currently using SMBG for managing their diabetes.
* Subject must be able to read and understand English
* In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
* Subject must have access to an internet connected computer for uploading data from the blood glucose meter and FreeStyle Libre system.
* Subject must be willing and able to provide written signed and dated informed consent.

Exclusion Criteria:

* Subject is a member of the Site Staff.
* Subject is currently using or has previously used a continuous glucose monitoring system for managing their diabetes
* Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
* Subject is pregnant or is attempting to become pregnant at the time of enrollment.
* Subject is on dialysis at the time of enrollment.
* Subject has concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff.
* Subject currently is participating in another clinical trial.
* Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects aged 18 years and older with type 1 or type 2 diabetes, who require daily blood glucose monitoring to manage their diabetes. At least 20% of the study population will be age 30 or below and 15% will be age 65 or older.
Sampling Method: Non-Probability Sample
Enrollment: 935 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Safety of the FreeStyle Libre Flash Glucose Monitoring System | Approximately one year per subject.
  The study is designed to characterize the safety of the FreeStyle Libre Flash Glucose Monitoring System when used in the intended study population.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care Inc
Locations (10):
- United States (10):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Baptist Diabetes Associates, P.A, Miami, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Iowa Diabetes & Endocrinology Research Center, Des Moines, Iowa
  - MassResearch, LLC, Waltham, Massachusetts
  - Henry Ford Medical Center, Detroit, Michigan
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - Texas Diabetes & Endocrinology, Round Rock, Texas
  - Clinical Trials of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No